CLINICAL TRIAL: NCT02565147
Title: Bivalirudin Infusion for Ventricular Infarction Limitation
Acronym: BIVAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility at the interim analysis.
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDCO-BIV-12-02; 2012-002314-39 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2015-10-01 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI, infarct size, CMR, bivalirudin
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint was evaluated by a core lab totally blinded to clinical information and the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPCI with Bivalirudin (Experimental): Bivalirudin was administered as a bolus (0.75 mg/kg) and an infusion (1.75 mg/kg/h) for the duration of the PPCI and continued for the first 4 h after completion of the procedure.
  Interventions: Procedure: PPCI; Drug: Bivalirudin
- PPCI with Heparin (Active Comparator): UFH was administered as a bolus according to standard of care for completion of PPCI per site. An ACT ≥250 s at the end of the procedure was recommended.
  Interventions: Procedure: PPCI; Drug: Heparin

INTERVENTIONS:
Procedure: PPCI — PPCI for treatment of participants presenting with large STEMI.
Drug: Bivalirudin — Bivalirudin is an anticoagulant that binds thrombin in a bivalent and reversible fashion and directly inhibits it.
  Other Names: Angiomax; Angiox
  Arms: PPCI with Bivalirudin
Drug: Heparin — Heparin is an anticoagulant.
  Other Names: UFH
  Arms: PPCI with Heparin

SUMMARY:
The purpose of this study is to evaluate whether the use of bivalirudin will reduce extent of the damage done to the heart muscle in participants who suffered a heart attack, compared to the comparator treatment (heparin).

DETAILED DESCRIPTION:
The study will assess the effect of bivalirudin administration during primary percutaneous coronary intervention (PPCI) and for 4 hours (h) afterwards, looking at contrast enhanced cardiac magnetic resonance imaging (CMR) assessed infarct size and on circulating markers of thrombosis and cell injury in participants treated with PPCI for a large myocardial infarction (MI).

The objective of this study is to determine whether bivalirudin, compared to heparin [unfractionated heparin (UFH)], for PPCI in large ST segment elevation myocardial infarction (STEMI) can:

Primary Objective • Reduce infarct size assessed by CMR 5 days (defined as 5 days ±72 h from randomisation) after PPCI

Secondary Objectives of this study are to determine the effects of bivalirudin compared with UFH treatment for PPCI in STEMI on:

* Other CMR derived parameters of myocardial recovery 5 days after PPCI (that is, left ventricular ejection fraction [LVEF], myocardial salvage index [MSI], and micro-vascular obstruction [MVO])
* LVEF by CMR at 90 days
* Modulate markers of thrombin activity and cell injury after reperfusion
* Coronary flow and micro-circulation at the end of PPCI
* Survival at 90 days

Approximately 200 participants will be randomized. Participants will be stratified prior to randomization: (a) according to total duration of ischemic pain (<6 h versus ≥6 h); (b) by site.

Diagnosis and Main Criteria for Selection: Adult participants (≥18 years) with an onset of ischemic symptoms of >20 minutes (min) and <12 h; a diagnosis of STEMI with ST segment elevation of ≥1 millimeter (mm) in ≥2 contiguous precordial leads, or presumably new left bundle branch block; had thrombolysis in myocardial infarction (TIMI) 0 or 1 flow in the infarct related artery (IRA); fulfilled angiographic criteria/score for a large infarction; and were candidates for PPCI will be enrolled. All participants should receive as soon as logistically feasible: aspirin (150-325 milligrams [mg] orally or 250-500 mg intravenously [IV]) and a loading dose of any approved P2Y12 inhibitor unless already on maintenance dose.

Bivalirudin will be administered at the time of PPCI at the approved dose of 0.75 mg/kilogram (kg) bolus followed by a 1.75 mg/kg/h infusion that will continue for 4 h after the completion of the index procedure.

Participants randomized to UFH should be treated according to the standard institutional protocol (including the timing and dosing of the UFH bolus). A target activated clotting time (ACT) of ≥250 seconds (s) was recommended.

Criteria for Evaluation:

Primary Endpoint:

• Infarct size assessed by CMR 5 days post-PPCI

Secondary Endpoints:

* CMR MVO assessment at 5 days
* CMR MSI at 5 days
* CMR assessment of LVEF at 5 days
* CMR assessment of LVEF at 90 days
* TIMI flow and Myocardial Blush Grade at end of PPCI
* In-hospital net adverse clinical events up to 5 days or discharge, whichever comes first (death, re-infarction, ischaemia driven revascularization, and Bleeding Academic Research Consortium ≥3 bleeding)
* Death at 90 days

Exploratory assessments:

• Assess patterns between comparator groups at various peri-procedural time points with respect to but not limited to: micro-particle release, thrombin anti thrombin complexes, myeloperoxidase

Sub-study:

• Index microcirculatory resistance

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Experienced ischemic symptoms of >20 min and <12 h and had a diagnosis of STEMI with ST segment elevation of ≥1 mm in ≥2 contiguous precordial leads, or presumably new left bundle branch block
3. Provided written informed consent or witnessed consent in countries and sites where such participant consenting is applicable, before initiation of any study-related procedures
4. Had TIMI 0 or 1 flow in the IRA on initial angiogram
5. Fulfilled angiographic criteria/score for a large infarction based on initial angiogram (Alberta Provincial Project for Outcome Assessment in Coronary Heart Disease score of ≥21)
6. Were candidates for PPCI
7. Administration of an initial dose of 150 to 325 mg orally (or 250 to 500 mg IV) and a loading dose of any approved P2Y12 inhibitor

Exclusion Criteria:

1. Contraindication or known hypersensitivity to bivalirudin or UFH
2. Refusal to receive blood transfusion/products
3. Participants requiring staged coronary artery bypass graft procedure within the first 90 days
4. Known international normalized ratio ≥2 or known prothrombin time >1.5 times upper limit of normal on the day of the index PPCI, or known history of bleeding diathesis
5. Therapy with vitamin K antagonists within 72 h of PPCI
6. Therapy with dabigatran, rivaroxaban, or other oral anti-Xa or antithrombin agents within 48 h of PPCI
7. History of hemorrhagic stroke, intracranial hemorrhage, intracerebral mass, aneurysm, arteriovenous malformation, or recent head injury (within the last 5 days)
8. Participants with previous history of Q-wave MI
9. Known glomerular filtration rate (GFR) <30 milliliter/min or dialysis dependent
10. Major surgery within the previous 30 days
11. Minor surgery/biopsy exclusions in the past 3 days
12. Upper gastrointestinal or genitourinary bleed 30 days prior to randomization
13. Stroke or transient ischemic attack 30 days prior to randomization
14. Administration of thrombolytics or glycoprotein IIb/IIIa inhibitor 72 h prior to PPCI
15. Administration of enoxaparin 8 h prior to PPCI
16. Administration of bivalirudin 12 h prior to PPCI
17. Administration of fondaparinux or other low molecular weight heparin 24 h prior to PPCI
18. Known contraindications to aspirin or P2Y12 inhibitors
19. Known allergy that cannot be pre-medicated to iodinated contrast
20. Known contraindication to CMR
21. Women of child bearing potential (see below)
22. Previous enrollment (participants are considered enrolled upon Randomization) in this study
23. Treatment with other investigational drugs or devices within the 30 days preceding enrollment or planned use of other investigational drugs or devices before the primary endpoint of this study had been reached
24. Participants with a body weight >150 kg

Child bearing potential was defined as:

A female participant was considered to have childbearing potential unless she met at least 1 of the following criteria:

* Age ≥50 years and naturally amenorrheic for ≥1 year (amenorrhea following cancer therapy did not rule out childbearing potential)
* Premature ovarian failure confirmed by a specialist gynecologist
* Previous bilateral salpingo-oophorectomy or hysterectomy
* XY genotype, Turner's syndrome, uterine agenesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Van Geuns, MD, Principal Investigator — Thorax Centrum, Erasmus Medisch Centrum, s-Grave dijkwal 230, 3015 CE Rotterdam, the Netherlands; Ludovic Drouet, MD, Principal Investigator — Hospital Lariboisiere, Angio-Hematologie, 2 Rue Ambroise Pare, 75475 Paris Cedex 10, France
Locations (4):
- France (2):
  - Hopital Ambroise Paré, Boulogne
  - Hospital Lariboisière, Paris
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Alderman EL, Stadius M. The angiographic definitions of the Bypass Angioplasty Revascularization Investigation. Coronary Artery Disease 1992;3: 1189-1207
- [Background] Graham MM, Faris PD, Ghali WA, Galbraith PD, Norris CM, Badry JT, Mitchell LB, Curtis MJ, Knudtson ML; APPROACH Investigators (Alberta Provincial Project for Outcome Assessment in Coronary Heart Disease. Validation of three myocardial jeopardy scores in a population-based cardiac catheterization cohort. Am Heart J. 2001 Aug;142(2):254-61. doi: 10.1067/mhj.2001.116481. PMID 11479464
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Background] Lowe JE, Reimer KA, Jennings RB. Experimental infarct size as a function of the amount of myocardium at risk. Am J Pathol. 1978 Feb;90(2):363-79. PMID 623206
- [Background] Ortiz-Perez JT, Meyers SN, Lee DC, Kansal P, Klocke FJ, Holly TA, Davidson CJ, Bonow RO, Wu E. Angiographic estimates of myocardium at risk during acute myocardial infarction: validation study using cardiac magnetic resonance imaging. Eur Heart J. 2007 Jul;28(14):1750-8. doi: 10.1093/eurheartj/ehm212. Epub 2007 Jun 22. PMID 17586811
- [Background] Reimer KA, Ideker RE, Jennings RB. Effect of coronary occlusion site on ischaemic bed size and collateral blood flow in dogs. Cardiovasc Res. 1981 Nov;15(11):668-74. doi: 10.1093/cvr/15.11.668. PMID 7326685
- [Background] Seiler C, Kirkeeide RL, Gould KL. Basic structure-function relations of the epicardial coronary vascular tree. Basis of quantitative coronary arteriography for diffuse coronary artery disease. Circulation. 1992 Jun;85(6):1987-2003. doi: 10.1161/01.cir.85.6.1987. PMID 1591819
- [Background] Seiler C, Kirkeeide RL, Gould KL. Measurement from arteriograms of regional myocardial bed size distal to any point in the coronary vascular tree for assessing anatomic area at risk. J Am Coll Cardiol. 1993 Mar 1;21(3):783-97. doi: 10.1016/0735-1097(93)90113-f. PMID 8436762
- [Background] Wu E, Judd RM, Vargas JD, Klocke FJ, Bonow RO, Kim RJ. Visualisation of presence, location, and transmural extent of healed Q-wave and non-Q-wave myocardial infarction. Lancet. 2001 Jan 6;357(9249):21-8. doi: 10.1016/S0140-6736(00)03567-4. PMID 11197356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants who underwent successful primary percutaneous coronary intervention (PPCI) defined as thrombolysis in myocardial infarction (TIMI) Flow of 2 or 3, underwent cardiac magnetic resonance imaging (CMR) at 5 days, and were without major protocol deviations were included in the per-protocol population (primary/secondary analyses).
Groups:
- PPCI With Bivalirudin: Bivalirudin was administered as a bolus (0.75 milligrams [mg]/kilogram [kg]) and an infusion (1.75 mg/kg/hours [h]) for the duration of the PPCI and continued for the first 4 h after completion of the procedure.
- PPCI With Heparin: Unfractionated heparin (UFH) was administered as a bolus according to standard of care for completion of PPCI per site. An activated clotting time (ACT) ≥250 seconds (s) at the end of the procedure was recommended.
Period: Overall Study
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Started | 38 | 40
Received Study Drug (Safety Population included all enrolled participants who received either bivalirudin or UFH.) | 38 | 40
Per-Protocol Population (Enrolled participants who underwent successful PPCI and Day-5 CMR without major protocol deviations.) | 28 | 36
Completed | 32 | 37
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled participants who received either bivalirudin or UFH.
Groups:
- Total: Total of all reporting groups
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (11.4) | 61.2 (13.2) | 62.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 28 | 34 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 21 | 22 | 43
  France | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: CMR Assessment Of Infarct Size At Day 5
Description: Size of cardiac infarct, expressed as grams, as assessed by CMR. The use of CMR has dramatically improved the ability for accurate infarct size estimations and is therefore currently considered the gold standard. The number of participants and their mean reported infarct size, as grams, at Day 5 are presented.
Time Frame: 5 days post PPCI
Population: All enrolled participants who underwent successful PPCI and CMR without major protocol deviations (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Grams | 25.0 (19.7) | 27.1 (20.7)
Statistical Analysis 1: Comparison: PPCI With Bivalirudin vs PPCI With Heparin; Test type: Superiority; p = 0.7505, Wilcoxon Rank Sum Test

2. Secondary Outcome: CMR Assessment Of Myocardial Salvage Index (MSI) At Day 5
Description: MSI is a CMR-derived parameter of myocardial recovery and treatment efficacy that allows comparisons among infarcts of different sizes. MSI is calculated as the difference between the area at risk (AAR) and the final infarct size, divided by the AAR, and it is expressed as a percentage of AAR. An MSI of 100% indicates maximum treatment success, whereas an MSI of 0% indicates no treatment benefit. The number of participants and their mean-reported MSI at Day 5 are presented.
Time Frame: 5 days post PPCI
Population: All enrolled participants who underwent successful PPCI and CMR without major protocol deviations (Per-Protocol Population) and participants with a successful CMR assessment of MSI.
Measure: Mean (Standard Deviation); unit: Percentage of AAR
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 12 | 15
Percentage of AAR | 39.4 (19.3) | 51.2 (21.7)

3. Secondary Outcome: CMR Assessment Of Micro-vascular Obstruction (MVO) At Day 5
Description: Early and late assessment of MVO, expressed as grams, as assessed by CMR. MVO is an established complication of coronary reperfusion therapy for acute myocardial infarction. MVO occurs in the setting of reperfusion following prolonged myocardial ischemia and provides incremental prognostic information beyond infarct size, to which it is related. Early MVO is a prolonged (approximately 60 s) perfusion deficit in dynamic gadolinium (Gd) first-pass images that is determined within 2 minutes (min) of administration of the Gd-based contrast agent. Late MVO is usually assessed as a hypointense infarct core on late-Gd-enhancement images acquired 10 min after contrast administration.
  The number of participants and their mean reported early and late MVO, as grams, at Day 5 are presented.
Time Frame: 5 days post PPCI
Population: All enrolled participants who underwent successful PPCI and CMR without major protocol deviations (Per-Protocol Population) and participants with a successful CMR assessment of MVO.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Grams
  CMR Early MVO Assessment: number analyzed (Participants) | 23 | 28
  CMR Early MVO Assessment | 5.3 (5.8) | 7.7 (6.3)
  CMR Late MVO Assessment: number analyzed (Participants) | 27 | 35
  CMR Late MVO Assessment | 3.7 (5.7) | 4.2 (4.5)

4. Secondary Outcome: CMR Assessment Of Left Ventricular Ejection Fraction (LVEF) At Day 5
Description: Percentage of cardiac LVEF as assessed by CMR. LVEF is a measurement of the percentage of blood ejected out of the left ventricle with each contraction. The number of participants and their mean reported LVEF, as a percentage of blood, at Day 5 are presented.
Time Frame: 5 days post PPCI
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Blood
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Percentage of Blood | 48.5 (11.0) | 48.6 (10.9)

5. Secondary Outcome: CMR Assessment Of LVEF At Day 90
Description: Percentage of cardiac LVEF as assessed by CMR. LVEF is a measurement of the percentage of blood ejected out of the left ventricle with each contraction. The number of participants and their mean reported LVEF, as a percentage of blood, at Day 90 are presented.
Time Frame: 90 days post PPCI
Population: All enrolled participants who underwent successful PPCI and CMR without major protocol deviations (Per-Protocol Population) and participants with a successful CMR assessment of LVEF at Day 90.
Measure: Mean (Standard Deviation); unit: Percentage of Blood
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 22 | 29
Percentage of Blood | 54.6 (12.0) | 49.1 (12.1)

6. Secondary Outcome: TIMI Flow And Myocardial Blush Grade (MBG) At End Of PPCI
Description: TIMI flow (grade 0-3) is an angiographic determination of briskness of epicardial coronary blood flow: TIMI 0 flow (no perfusion); TIMI 1 flow (penetration without perfusion); TIMI 2 flow (partial reperfusion); TIMI 3 flow (complete perfusion/normal flow).
  MBG (grade 0-3) is an angiographic method for determination of blood flow in the distal myocardial vascular bed. Blush grades: 0 = failure of dye to enter the micro-vasculature; 1 = dye slowly enters but fails to exit the micro-vasculature; 2 = delayed entry and exit of dye from the micro-vasculature; 3 = normal entry and exit of dye from the micro-vasculature. Blush that is only mildly intense throughout the washout phase, but fades minimally, is also classified as grade 3.
  The number of participants and their mean reported TIMI flow and MBG grades at the end of PPCI are presented.
Time Frame: 1 day (end of PPCI)
Population: All enrolled participants who underwent successful PPCI and CMR without major protocol deviations (Per-Protocol Population) and participants with a detectable TIMI Flow and MBG at the end of PPCI.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Units on a Scale
  TIMI Flow Grade | 2.8 (0.4) | 2.8 (0.4)
  MBG: number analyzed (Participants) | 22 | 29
  MBG | 1.8 (1.2) | 1.5 (1.2)

7. Secondary Outcome: Percentage of Participants With In-Hospital Net Adverse Cardiac Events (NACE) At Day 5
Description: The NACE at 5 days is the composite of major bleeding (Bleeding Academic Research Consortium Type 3 or greater [BARC type ≥3]), death, re-infarction, and ischaemia driven revascularization (IDR).
  In brief, BARC ≥3 includes: Type 3a-3c, clinical, laboratory, and/or imaging evidence of bleeding; Type 4, coronary artery bypass grafting-related bleeding; Type 5, fatal bleeding that directly results in death that is either clinically suspicious or is confirmed as the cause of death.
  A participant was defined to have a composite event if the participant experienced at least 1 of the components. If the participant did not have any of the components, then he or she did not have the composite endpoint. If a participant had more than 1 of the components, he or she was only counted once in the determination of the total number of participants experiencing the composite endpoint.
  The percentage of participants with in-hospital NACE up to Day 5 is presented.
Time Frame: 5 days post PPCI or at discharge, whichever occurs first
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Percentage of Participants | 7.1 | 8.3

8. Secondary Outcome: Death At Day 90
Description: Participant survival during the clinical follow-up period is presented as the number of participants with reported death at 90 days post PPCI.
Time Frame: 90 days post PPCI
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 28 | 36
Participants | 0 | 1

9. Other Pre Specified Outcome: Index Of Microcirculatory Resistance (IMR)
Description: IMR, a predictor of clinical outcome, is a readily available, quantitative, and reproducible method for invasively assessing coronary microvascular function. It is measured using the thermodilution technique and defined as mean distal coronary pressure, expressed in millimeters (mm) of mercury (Hg), multiplied by the mean hyperemic transit time (s) (mmHg*s). Higher IMR values indicate poorer microcirculation and are associated with a worse clinical outcome. A cutoff point of 32 (associated with better clinical outcomes) was selected as the threshold. Only participants at study locations with previous experience in IMR measurements participated in this sub study.
  The number of participants and their mean reported IMR at the end of PPCI are presented.
Time Frame: 1 day (end of PPCI)
Population: All participants enrolled into the randomized trial (Intent-to-treat [ITT] Population) who took part in the IMR sub study (IMR-ITT).
Measure: Mean (Standard Deviation); unit: mmHg*s
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
Number analyzed (Participants) | 25 | 25
mmHg*s | 43.49 (21.62) | 68.66 (35.77)

ADVERSE EVENTS:
Time Frame: Up to 5 days (±36 h) post randomization/discharge
Arm/Group | PPCI With Bivalirudin | PPCI With Heparin
All-Cause Mortality (participants affected / at risk) | 1/38 | 1/40
Serious Adverse Events (participants affected / at risk) | 6/38 | 7/40
Other Adverse Events (participants affected / at risk) | 11/38 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PPCI With Bivalirudin (N=38) | PPCI With Heparin (N=40)
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 0
Coronary artery perforation (Cardiac disorders) | 1 | 0
Myocardial rupture (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PPCI With Bivalirudin (N=38) | PPCI With Heparin (N=40)
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Since the measured difference in infarct size at Day 5 (by CMR) was <18%, the study was terminated for futility at the interim analysis as pre-defined in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days